CLINICAL TRIAL: NCT01184391
Title: Single-Dose Fasting Bioequivalence Study of Divalproex Sodium Delayed-Release Tablets (500 mg; Mylan) and Depakote Tablets (500 mg; Abbott) in Healthy Adult Male And Female (Not of Childbearing Potential) Volunteers
Brief Title: Bioequivalence Study of Divalproex Sodium Delayed-Release Tablets, 500 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Vice President, Regulatory Affairs, Mylan Pharmaceuticals Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DIVA-0771
Record Dates: First submitted 2009-09-24; First posted 2010-08-18 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
MeSH Terms: interventions — Valproic Acid

ARMS (2):
- Test: Divalproex Sodium (Experimental): DIVALPROEX SODIUM DELAYED-RELEASE TABLETS, USP, 500 MG
  Interventions: Drug: DIVALPROEX SODIUM DELAYED-RELEASE TABLETS, USP, 500 MG
- Reference: Depakote Tablets (Active Comparator): DEPAKOTE® Tablets, 500 MG Abbott Laboratories
  Interventions: Drug: DEPAKOTE® Tablets, 500 MG

INTERVENTIONS:
Drug: DEPAKOTE® Tablets, 500 MG — 1 x 500 mg tablet, under fasting conditions
  Arms: Reference: Depakote Tablets
Drug: DIVALPROEX SODIUM DELAYED-RELEASE TABLETS, USP, 500 MG — 1 X 500 mg Tablet, under fasting conditions.
  Arms: Test: Divalproex Sodium

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's divalproex sodium-delayed-release tablets 500 mg tablets to Abbott's Depakote® 500 mg tablets following a single, oral 500 mg (1 x 500 mg) dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Females not of child bearing potential and males.

   * No hormonal contraceptives or hormonal replacement therapies are permitted in this study.
   * Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

     * postmenopausal with spontaneous amenorrhea for at least one (1) year, or spontaneous amenorrhea for less than one (1) year with serum FSH levels > 40 mIU/ml, or
     * bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
     * total hysterectomy and an absence of bleeding for at least 3 months.
   * During the course of the study, from study screen until study exit - including the washout period, all men must use a spermicide containing barrier method of contraception in addition to their current contraceptive method. These instructions should be documented in the informed consent form.
3. Weight Restrictions:

   * At least 60 kg (132 lbs) for men and
   * At least 48 kg (106 lbs) for women
   * All subjects will have a Body Mass Index (BMI) less than or equal to 30 but greater than or equal to 19 (see Part II, Administrative Aspects of Bioequivalence Protocols). BMI values should be rounded to the nearest integer (ex. 30.4 rounds down to 30, while 18.5 rounds up to 19)
4. All subjects should be judged by the principal or sub-investigator physician listed on the Form FDA 1572 as normal and healthy during a pre-study medical evaluation performed within 21 days of the initial dose of study medication which will include:
5. Normal or non-clinically significant physical examination including vital signs,
6. Within normal limits or non-clinically significant laboratory evaluation results for the following tests:

   * Serum Chemistries: sodium, potassium, chloride, BUN, iron, albumin, total protein AST, Alk. Phos., Calcium, Creatinine, ALT, Total bilirubin, Total Cholesterol, Phosphate, Uric Acid, Non-fasting Glucose Triglycerides
   * Hematology: Platelet Count, Hemoglobin, Leukocyte Differential, Hematocrit, Red Blood Cells
   * Urinalysis: Appearance, Specific Gravity, Protein pH, Microscopic Examination
7. Negative Hepatitis B and Hepatitis C tests,
8. Negative HIV test,
9. Normal or non-clinically significant 12-lead ECG
10. Negative urine drug screen for all of the following compounds: amphetamines, barbiturates, benzodiazepines, cannabinoid, cocaine, methadone, opiates, and phencyclidine

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   * Use of any tobacco-containing products within 1 year of the start of the study.
   * Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   * Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   * Any recent, significant change in dietary or exercise habits.
   * Individual has a history of drug and/or alcohol abuse.
3. Medications:

   * Use of any prescription or over-the-counter (OTC) medications within fourteen (14) days prior to the initial dose of study medication.
   * Use of any hormone replacement therapy within 3 months prior to study medication dosing.
   * Use of any medication known to induce or inhibit hepatic enzyme activity within 28 days prior to the initial dose of study medication (see Part II, Administrative Aspects of Bioequivalence Protocols for list).
4. Diseases:

   * History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, congenital metabolic disorders or neurologic disease.
   * Acute illness at the time of either the pre-study medical evaluation or dosing.
   * All laboratory values reflecting hepatic function must be with in 10% of the upper range of normal in order to be considered not clinically significant.
5. Subjects who have known urea cycle disorders which are a group of uncommon genetic abnormalities (e.g. ornithine transcarbamylase deficiency).
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to Divalproex Sodium or any related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Cmax | 30 days
  Maximum plasma concentration (micrograms/mL)
AUCL | 30 days
  Area under the concentration time curve from time zero to the last measurable concentration(micrograms x mL/hr)
AUCI | 30 days
  Area under the concentration time curve from time zero to infinity (micrograms x mL/hr)

CONTACTS AND LOCATIONS:
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc - Clinical Trial Results — http://www.mpibiostudies.com